CLINICAL TRIAL: NCT06671314
Title: Adoption of Novel Heart Failure Therapy and Outcomes in Patients With Heart Failure With Mildly Reduced or Preserved Ejection Fraction
Brief Title: Heart Failure Therapy and Outcomes in Patients With Heart Failure With Mildly Reduced or Preserved Ejection Fraction
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: CLCZ696DUS07
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Heart Failure Cohort: Adults hospitalized with heart failure from the Get With The Guidelines - Heart Failure (GWTG-HF) registry and enrolled in Medicare Fee-for-Service at the time of discharge. Patients had heart failure with preserved or mildly reduced ejection fraction.

SUMMARY:
This was a retrospective observational cohort study using patient data from the Get With The Guideline-Heart Failure (GWTG-HF) registry linked to Medicare Fee-for-Service (FFS) claims. The main goal of the study was to compare home-time in Medicare FFS patients with heart failure with mildly reduced or preserved ejection fraction discharged with sacubitril/valsartan versus those discharged without sacubitril/valsartan.

ELIGIBILITY:
Inclusion criteria:

* Hospitalized for heart failure from 01 January 2016 to 30 September 2021.
* Were discharged alive (any discharge disposition other than "Expired").
* Had Mildly reduced or preserved ejection fraction (41% to 60%).
* Had non-missing record of SAC/VAL use at discharge.
* Continuously enrolled in Medicare Part A & B for the 12 months following the index HF hospitalization discharge date or until death.

Exclusion criteria:

* Patients who left against medical advice (AMA), were transferred to an acute care facility, or discharged to hospice care.
* Patients who had dialysis as an in-hospital procedure.
* Patients with a medical history of chronic dialysis.
* Patients with an in-hospital procedure of heart transplantation.
* Patients with a medical history of heart transplantation.
* Patients with an in-hospital procedure of left ventricular assist device.
* Patients with a medical history of left ventricular assist device.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 42494 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Time Spent 30 Days Post-discharge by Discharge Sacubitril/Valsartan (SAC/VAL) Prescription Status | Post-discharge at Day 30
  Time spent included home-time days, hospital days, skilled nursing facility days, rehab days, other institutional days, and death days. Home-time was defined as the number of days alive and out of the hospital, skilled nursing facility or inpatient rehabilitation facility.
  SAC/VAL prescription status: with SAC/VAL prescription and without SAC/VAL prescription.
Time Spent 90 Days Post-discharge by Discharge SAC/VAL Prescription Status | Post-discharge at Day 90
  Time spent included home-time days, hospital days, skilled nursing facility days, rehab days, other institutional days, and death days. Home-time was defined as the number of days alive and out of the hospital, skilled nursing facility or inpatient rehabilitation facility.
  SAC/VAL prescription status: with SAC/VAL prescription and without SAC/VAL prescription.
Time Spent 180 Days Post-discharge by Discharge SAC/VAL Prescription Status | Post-discharge at Day 180
  Time spent included home-time days, hospital days, skilled nursing facility days, rehab days, other institutional days, and death days. Home-time was defined as the number of days alive and out of the hospital, skilled nursing facility or inpatient rehabilitation facility.
  SAC/VAL prescription status: with SAC/VAL prescription and without SAC/VAL prescription.
Time Spent 365 Days Post-discharge by Discharge SAC/VAL Prescription Status | Post-discharge at Day 365
  Time spent included home-time days, hospital days, skilled nursing facility days, rehab days, other institutional days, and death days. Home-time was defined as the number of days alive and out of the hospital, skilled nursing facility or inpatient rehabilitation facility.
  SAC/VAL prescription status: with SAC/VAL prescription and without SAC/VAL prescription.

SECONDARY OUTCOMES:
Number of All-cause Mortality Patients at 30, 90, 180, and 365 Days After Discharge With a Sacubitril/Valsartan (SAC/VAL) Prescription | Post-discharge at Days 30, 90, 180, and 365
Number of All-cause Mortality Patients at 30, 90, 180, and 365 Days After Discharge Without a SAC/VAL Prescription | Post-discharge at Days 30, 90, 180, and 365
Number of All-cause Mortality or Heart Failure (HF) Hospitalization Patients at 30, 90, 180, and 365 Days After Discharge With a SAC/VAL Prescription | Post-discharge at Days 30, 90, 180, and 365
Number of All-cause Mortality or HF Hospitalization Patients at 30, 90, 180, and 365 Days After Discharge Without a SAC/VAL Prescription | Post-discharge at Days 30, 90, 180, and 365
Number of All-cause Hospitalization Patients at 30, 90, 180, and 365 Days After Discharge With SAC/VAL Prescription | Post-discharge at Days 30, 90, 180, and 365
  All-cause hospitalization was defined as any inpatient claim for post-discharge admission to an acute care hospital excluding transfers and hospitalizations for rehabilitation.
Number of All-cause Hospitalization Patients at 30, 90, 180, and 365 Days After Discharge Without a SAC/VAL Prescription | Post-discharge at Days 30, 90, 180, and 365
  All-cause hospitalization was defined as any inpatient claim for post-discharge admission to an acute care hospital excluding transfers and hospitalizations for rehabilitation.
Number of Patients Hospitalized for HF at 30, 90, 180, and 365 Days After Discharge With a SAC/VAL Prescription | Post-discharge at Days 30, 90, 180, and 365
  HF hospitalization was defined as any inpatient claim with a primary diagnosis of HF (International Classification of Diseases, 10th revision, Clinical Modification [ICD-10-CM] diagnosis codes I098.1, I50.*, I11.0, I13.0, I13.2) excluding transfers.
Number of Patients Hospitalized for HF at 30, 90, 180, and 365 Days After Discharge Without a SAC/VAL Prescription | Post-discharge at Days 30, 90, 180, and 365
  HF hospitalization was defined as any inpatient claim with a primary diagnosis of HF (International Classification of Diseases, 10th revision, Clinical Modification [ICD-10-CM] diagnosis codes I098.1, I50.*, I11.0, I13.0, I13.2) excluding transfers.
Number Patients Hospitalized for Dialysis or End-Stage Kidney Disease at 365 Days After Discharge With and Without a SAC/VAL Prescription | Post-discharge at Day 365
  Hospitalization for dialysis or end-stage kidney disease was defined as any inpatient claim having a primary diagnosis of dialysis or end-stage kidney disease (International Classification of Diseases, 10th revision, Clinical Modification [ICD-10-CM] diagnosis codes Z99.2, Z49, N18.5, N18.6; or ICD.9 - 585.6, V45.11, V56.0, V56.8)
Number Patients Hospitalized for a Metabolic/Nutritional Disorder at 365 Days After Discharge With and Without a SAC/VAL Prescription | Post-discharge at Day 365
  Hospitalization for metabolic/nutritional reasons was defined as any inpatient claims with Diagnosis-related group (DRG) codes 640, 641.
Number Patients Hospitalized for Urinary Tract Infection at 365 Days After Discharge With and Without a SAC/VAL Prescription | Post-discharge at Day 365
  Hospitalization for urinary tract infection was defined as any inpatient claims with a primary diagnosis of International Classification of Diseases, 10th revision, Clinical Modification (ICD-10-CM) code N39.0.
Number Patients Hospitalized for a Hip Fracture at 365 Days After Discharge With and Without a SAC/VAL Prescription | Post-discharge at Day 365
  Hospitalization for hip fracture was defined as any inpatient claims with a primary diagnosis fracture of the neck of the femur.
Difference in Days of Home-time Between Discharge With and Without SAC/VAL Prescription | Post-discharge at Days 30, 90, 180, and 365
  Home-time was defined as the number of days alive and out of the hospital, skilled nursing facility or inpatient rehabilitation facility.
Difference in All-cause Mortality Between Discharge With and Without SAC/VAL Prescription | Post-discharge at Days 30, 90, 180, and 365
Difference in Composite Measure Between Discharge With and Without SAC/VAL Prescription | Post-discharge at Days 30, 90, 180, and 365
  Composite measure: all-cause mortality or heart failure hospitalization.
Difference in All-cause Re-hospitalization Between Discharge With and Without SAC/VAL Prescription | Post-discharge at Days 30, 90, 180, and 365
Difference in HF Re-hospitalization Between Discharge With and Without SAC/VAL Prescription | Post-discharge at Days 30, 90, 180, and 365
Difference in Hospitalization for Metabolic/Nutritional Disorder Between Discharge With and Without SAC/VAL Prescription | Post-discharge at Day 365
  Hospitalization for metabolic/nutritional reasons was defined as any inpatient claims with Diagnosis-related group (DRG) codes 640, 641.
Difference in Hospitalization for Urinary Tract Infection Between Discharge With and Without SAC/VAL Prescription | Post-discharge at Day 365
  Hospitalization for urinary tract infection was defined as any inpatient claims with a primary diagnosis of International Classification of Diseases, 10th revision, Clinical Modification (ICD-10-CM) code N39.0.
Difference in Hospitalization for Hip Fracture Between Discharge With and Without SAC/VAL Prescription | Post-discharge at Day 365
  Hospitalization for hip fracture was defined as any inpatient claims with a primary diagnosis fracture of the neck of the femur.
Number of All-cause Re-hospitalizations per Patient by Discharge SAC/VAL Prescription Status | Post-discharge at Day 365
  SAC/VAL prescription status: with SAC/VAL prescription and without SAC/VAL prescription.
Number of HF Re-hospitalizations per Patient by Discharge SAC/VAL Prescription Status | Post-discharge at Day 365
  SAC/VAL prescription status: with SAC/VAL prescription and without SAC/VAL prescription.
All-cause Re-hospitalization Length of Stay by Discharge SAC/VAL Prescription Status | Post-discharge at Day 365
  SAC/VAL prescription status: with SAC/VAL prescription and without SAC/VAL prescription.
All-cause HF-related Re-hospitalization Length of Stay by Discharge SAC/VAL Prescription Status | Post-discharge at Day 365
  SAC/VAL prescription status: with SAC/VAL prescription and without SAC/VAL prescription.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States